CLINICAL TRIAL: NCT00260897
Title: Molecular Genetic Study of Avascular Necrosis of the Femoral Head-Revealing ANFH Pathogenesis Mechanism by Cell and Animal Models
Brief Title: Molecular Genetic Study of Avascular Necrosis of the Femoral Head
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Other Study IDs: EC 9206002
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Osteonecrosis
Keywords: avascular necrosis of the femoral head; genotyping; linkage analysis; pathogenesis; therapy
MeSH Terms: conditions — Osteonecrosis; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Avascular necrosis of the femoral head (ANFH) is a debilitating disease that commonly leads to destruction of the hip joint in patients at middle age of life and often requires surgical intervention. Previously, we have identified the collagen type II, alpha 1 (COL2A1) gene as the ANFH disease gene. In this grant proposal, we will establish cell ine and animal models to understand the pathophysiology of ANFH, and extend our ongoing study for identifying genes responsible for non-familiar ANFH by looking into other interacting molecules of the pathway.

DETAILED DESCRIPTION:
Avascular necrosis of the femoral head (ANFH) is a debilitating disease that usually leads to destruction of the hip joint in the third to fifth decade of life (average age, 36 years). The disease prevalence is unknown, but it has been estimated that 10,000-20,000 new cases per year are diagnosed in the United State. Nearly half of the patients eventually require hip replacement before 40 years of age. The etiology of ANFH is unknown but previous studies indicated that heritable thrombophilia (increased tendency to form thrombi) and hypofibrinolysis (reduced ability to lyse thrombi), alcohol intake, and steroid use are risk factors for ANFH.

Although the majority of idiopathic ANFH cases are sporadic, recently we identified three ANFH families showing autosomal dominant inheritance. By genome-wide scan, a significant two-point LOD score of 3.45 at = 0 was obtained between one ANFH pedigree and marker D12S85 on chromosome 12. High-resolution mapping was conducted in a second ANFH family and replicated the linkage to D12S368. When an age-dependent penetrance model was applied, the combined multipoint LOD score achieved 6.43 between D12S1663 and D12S85. Furthermore, by using haplotype analysis and gene-based mutation detection, we have identified the collagen type II, alpha 1 (COL2A1) gene, as the ANFH disease gene. Re-sequencing of the type II collagen (COL2A1) gene demonstrated a glycine with serine mutation in the G-X-Y repeat of type II collagen, in all affected individuals in three pedigrees. In the Pedigree I, a 3665G >A mutation in exon 50 of the COL2A1 gene (Genbank accession number NM_001844) and the substitution resulted in a Gly1170Ser codon change (Genbank accession number NP_001835). A second pedigree was shown to harbor the same mutation but the mutant allele existed in a different haplotype background. In a third pedigree, a 2306G>A mutation occurred in exon 33 of the gene (Genbank accession number NM_001844), causing glycine to serine change at codon 717 (Genbank accession number NP_001835).

On this basis, we propose to study the pathophysiological mechanism(s) of inherited and sporadic ANFH. The main focus of this project includes: (1) Establishing cell line and animal models to investigate the molecular basis of ANFH pathogenesis. (2) Conducting genetic analysis on sporadic ANFH cases, including those who are idiopathic, alcohol consumers or steroid-induced. (3) Using COL2A1 gene as a target, we will design novel therapeutics and prediction procedures to improve the management of the ANFH patients.

ELIGIBILITY:
Inclusion Criteria:

- avascular necrosis of the femoral head

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2003-05; Study Completion 2008-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ming Chen, M.D., Principal Investigator — Department of Orthopaedics and Traumatology, Taipei Veterans General Hospital
Locations (1):
- Division of Molecular and Genomic Medicine, National Health Research Institutes, Miaoli County, Taiwan

REFERENCES:
- See also: Related Info — http://www.nhri.org.tw